CLINICAL TRIAL: NCT04288401
Title: Prevalence of Osteosarcopenic Obesity in Older Community-dwelling Adults in Turkey
Brief Title: Prevalence of Osteosarcopenic Obesity in Older Adults
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Goztepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Esma Nur KOLBAŞI, Principal Investigator, Istanbul Medeniyet University
Other Study IDs: IstanbulMU3
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Obesity; Sarcopenia; Osteopenia; Osteoporosis
MeSH Terms: conditions — Obesity; Sarcopenia; Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Osteosarcopenic Obesity (OSO) is a syndrome characterized by the loss of bone and muscle in addition to increase in the fat tissue as a result of aging process. It is the latest point of impairment in the bone,muscle and adipose tissue in older adults. OSO, as the name suggests, is the combination of three syndrome frequently encountered in the elderly: osteopenia/osteoporosis, sarcopenia and obesity. The aims of study are to determine the prevalence of OSO syndrome in community-dwelling adults of Turkey and determine the possible factors regarding risk of falling in this population

ELIGIBILITY:
Inclusion Criteria:

* Age of 65 or over
* Being had been examined for all the primary outcome measures (i.e. the results of primary outcomes must be in the patient's file)

Exclusion Criteria:

* Severe cognitive dysfunction
* not being able to walk independently for 4 m

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: older adults at the age of 65 or over
Sampling Method: Non-Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
T score | 1 hour
  T scores of spine and femur neck examined with Dual X-Ray Absorptiometry. A T score<-2,5 will be classified as osteoporosis while a T score between -1 and -2,5 will be counted as osteopenia
Muscle Strength | 5 minutes
  Measured by hand held dynamometer. The cut-off scores for man and woman are 27 kg and 16 kg, respectively
Muscle Mass | 2 minutes
  Measured by bioimpedance analysis using Tanita TBF300. The cut-off scores for man and woman are 9,2 kg/m2 and 7,4 kg/m2, respectively
Muscle Performance | 3 minutes
  Tested by 4 meter walk test. If the gait speed is lower than 0,8 m/s, the test is positive.
Obesity | 2 minutes
  The fat percentage and the Body Mass Index measured by bioimpedance analysis using Tanita TBF300 is recorded. For BMI, 30 kg/m2 and over is classified as obesity whereas fat percentage of %35 and %28 (woman and man, respectively) and over was classified as obese.

SECONDARY OUTCOMES:
Comorbidity | 3 minutes
  Using Charlson Comorbidity Index
History of falls | 1 minutes
  A patient's self stated history of falls will be considered as having a history of fall or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Goztepe Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kolbasi EN, Demirdag F. Prevalence of osteosarcopenic obesity in community-dwelling older adults: a cross-sectional retrospective study. Arch Osteoporos. 2020 Oct 20;15(1):166. doi: 10.1007/s11657-020-00829-x. PMID 33079259